CLINICAL TRIAL: NCT06559657
Title: Investigation of the Compatibility Among Innovative Methods in Measuring the Area and Depth of Pressure Injuries
Brief Title: Investigation of the Consistency Between Innovative Methods for Measuring the Area and Depth of Pressure Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gul SAHBUDAK, Research assistant at the Department of Nursing Principles, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Nursing Faculty
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Pressure Injury; Innovativeness; Wound
Keywords: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wound area and depth measurement (Experimental): The area of the pressure injuries was measured using digital planimetry, the imitoMeasure mobile application, and the three-dimensional wound measurement method. Depth was measured using a sterile cotton swab and the three-dimensional wound measurement method.
  Interventions: Device: eKare Insight, imitoMeasure Mobile App, Visitrak

INTERVENTIONS:
Device: eKare Insight, imitoMeasure Mobile App, Visitrak — The wound size of the patients was measured with three different methods. Wound depth was measured using manual method and three-dimensional imaging devices.

SUMMARY:
Wound healing is a complex process and wound care and evaluation is one of the most important problems in current medicine. Wounds are seen in clinics as diabetic foot ulcers (DFU), arterial and venous ulcers, pressure injuries, surgical wounds and so on. Pressure injuries (PI) have a high mortality rate (29%) among elderly individuals. The prevalence of PIs in different countries worldwide varies between 6% and 18.5% in acute care settings. Wound assessment is an integral part of nursing practice.

Improper assessment of wounds may lead to inadequate wound care, resulting in delayed wound healing, increased risk of infection, increased costs, and decreased patient quality of life. Wound measurement is a useful quantitative finding in wound assessment, used as a practical approach to monitor wound healing. An ideal wound measurement method should be practical, comfortable for the patient, high accuracy, reliability and applicability. In clinical practice, it is essential to regularly reassess wounds to monitor changes in size, depth, and appearance over time.

With the emergence of new techniques and technologies, there is a need for methods that can be considered as the gold standard in the measurement of wound dimensions. It is seen in the literature that studies comparing two- and three-dimensional measurement methods are generally carried out on superficial wounds and very limited wound types. In addition, there are hardly any studies comparing depth measurements with three-dimensional methods. In this direction, it was necessary to conduct this study in order to create evidence-based data in the field. The research has the quality of being the first and original study in our country that evaluates the compatibility of innovative methods in the area measurement of PIs and measures the wound depth.

DETAILED DESCRIPTION:
Hypotheses H1: There is concordance between digital planimetry and the imitoMeasure mobile application in measuring wound area.

H2: There is concordance between digital planimetry and three-dimensional wound area measurement in measuring wound area.

H3: There is concordance between the imitoMeasure mobile application and three-dimensional wound area measurement in measuring wound area.

H4: There is concordance between measurement with a sterile cotton swab and three-dimensional wound measurement in assessing wound depth.

Aim: The aim of this study is to examine the concordance between digital planimetry, the imitoMeasure mobile application, and three-dimensional wound measurement methods in measuring the area of pressure injuries, and to compare the measurement of wound depth using a sterile swab with the three-dimensional wound measurement method.

Research Place and Time: This study was conducted between April 2022 and April 2024 in the intensive care unit of the Department of Anesthesiology and Reanimation at Ege University Medical Faculty Hospital.

Data Collection:

For the purpose of data collection in this study, the following were used: the "Individual and Wound Identification Form," the "Informed Consent Form," the "Digital Planimetry Device (Visitrak™)," the "Smith & Nephew Opsite Flexigrid Transparent Wound Dressing," the "imitoMeasure mobile application (iPhone 13)," the "eKare inSight device," and a "Sterile Cotton Swab."

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Volunteering to participate in research,
* Having at least Stage 2 pressure injury

Exclusion Criteria:

* Having Stage 1 pressure injuries
* Having a wound with a shape that makes 2D area measurement impossible
* Patients who cannot remain in the same position for a long time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Wound area measurment | Approximately 5 minutes until the wound is selected and the measurement is completed.
  It is the measurement of wound area with three different methods.
Wound depth measurment | Approximately 5 minutes until the wound is selected and the measurement is completed.
  It is the measurement of wound depth with two different methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Magny E, Vallet H, Cohen-Bittan J, Raux M, Meziere A, Verny M, Riou B, Khiami F, Boddaert J. Pressure ulcers are associated with 6-month mortality in elderly patients with hip fracture managed in orthogeriatric care pathway. Arch Osteoporos. 2017 Aug 29;12(1):77. doi: 10.1007/s11657-017-0365-9. PMID 28852954
- [Result] Anisuzzaman DM, Wang C, Rostami B, Gopalakrishnan S, Niezgoda J, Yu Z. Image-Based Artificial Intelligence in Wound Assessment: A Systematic Review. Adv Wound Care (New Rochelle). 2022 Dec;11(12):687-709. doi: 10.1089/wound.2021.0091. Epub 2021 Dec 20. PMID 34544270
- [Result] Tervo-Heikkinen TA, Heikkila A, Koivunen M, Kortteisto TR, Peltokoski J, Salmela S, Sankelo M, Ylitormanen TS, Junttila K. Pressure injury prevalence and incidence in acute inpatient care and related risk factors: A cross-sectional national study. Int Wound J. 2022 May;19(4):919-931. doi: 10.1111/iwj.13692. Epub 2021 Oct 4. PMID 34605185
- [Result] Tubaishat A, Papanikolaou P, Anthony D, Habiballah L. Pressure Ulcers Prevalence in the Acute Care Setting: A Systematic Review, 2000-2015. Clin Nurs Res. 2018 Jul;27(6):643-659. doi: 10.1177/1054773817705541. Epub 2017 Apr 27. PMID 28447852
- [Result] Little C, McDonald J, Jenkins MG, McCarron P. An overview of techniques used to measure wound area and volume. J Wound Care. 2009 Jun;18(6):250-3. doi: 10.12968/jowc.2009.18.6.42804. PMID 19661849
- [Result] Khong PCB, Yeo MSW, Goh CC. Evaluating an iPad app in measuring wound dimension: a pilot study. J Wound Care. 2017 Dec 2;26(12):752-760. doi: 10.12968/jowc.2017.26.12.752. PMID 29244972
- [Result] Keast DH, Bowering CK, Evans AW, Mackean GL, Burrows C, D'Souza L. MEASURE: A proposed assessment framework for developing best practice recommendations for wound assessment. Wound Repair Regen. 2004 May-Jun;12(3 Suppl):S1-17. doi: 10.1111/j.1067-1927.2004.0123S1.x. PMID 15230830
- [Result] Pena G, Kuang B, Szpak Z, Cowled P, Dawson J, Fitridge R. Evaluation of a Novel Three-Dimensional Wound Measurement Device for Assessment of Diabetic Foot Ulcers. Adv Wound Care (New Rochelle). 2020 Nov;9(11):623-631. doi: 10.1089/wound.2019.0965. Epub 2019 Oct 23. PMID 33095125
- [Derived] Sahbudak G, Gunes U. Comparing Digital, Mobile and Three-Dimensional Methods in Pressure Injury Measurement: Agreement in Surface Area and Depth Assessments. J Clin Nurs. 2026 Jan;35(1):172-181. doi: 10.1111/jocn.17813. Epub 2025 May 9. PMID 40346762